CLINICAL TRIAL: NCT00768612
Title: A Randomized, Double-Blind, Risperidone-Reference, Parallel-Group, Safety, and Tolerability Study of Vabicaserin (SCA-136) in Japanese Subjects With Acute Exacerbation of Schizophrenia
Brief Title: Study Evaluating Safety and Tolerability of Vabicaserin in Patients With Sudden Worsening of Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3153B1-2208
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Acute, Schizophrenia, Phase2a, Vabicaserin
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Lowest dose
  Interventions: Drug: SCA-136 50mg/day
- 2 (Experimental): Middle dose
  Interventions: Drug: SCA-136 150 mg/day
- 3 (Experimental): Highest dose
  Interventions: Drug: SCA-136 300mg/day
- 4 (Active Comparator): Positive Control
  Interventions: Drug: Risperidone 4mg/day

INTERVENTIONS:
Drug: SCA-136 50mg/day
  Arms: 1
Drug: SCA-136 150 mg/day
  Arms: 2
Drug: SCA-136 300mg/day
  Arms: 3
Drug: Risperidone 4mg/day
  Arms: 4

SUMMARY:
This study will evaluate the clinical safety and tolerability of vabicaserin in Japanese subjects that have a sudden worsening of their symptoms of schizophrenia. The study will also assess the efficacy of vabicaserin and compare it to risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between >=20 and =<65 years of age
* Current diagnosis and DSM-IV-TR diagnosis of schizophrenia type (295.10, 295.30 and 295.90)
* Total PANSS score >=70 and =< 120

Exclusion Criteria:

* Subjects who are hospitalized against their will
* Current Axis I primary psychiatric diagnosis other than schizophrenia
* A score of 3 on CDSS question 8 which pertains to suicide

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale PANSS | 6 week

SECONDARY OUTCOMES:
Calgary Depression Scale for Schizophrenia CDSS | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer